CLINICAL TRIAL: NCT00305292
Title: "Modafinil-Alcohol Interactions Assessed Using Tests of Thermal Stimulation, Cognition, Mood, and Motor Function in Healthy Volunteers"
Brief Title: Modafinil-Alcohol Interactions in Healthy Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study should be terminated as the study closed prior to 2007 and the investigator has since retired. No records are available.
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: H5612-27941-01
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Alcohol
MeSH Terms: interventions — Modafinil; Ethanol; Drug Interactions

INTERVENTIONS:
Drug: Modafinil-Alcohol Interactions

SUMMARY:
The UCSF Pain Clinical Research Center (PCRC) is conducting a study of the effects of modafinil (Provigil®; Vigiver, Alertec), alcohol and the combination on alertness, mood, visual motor and cognitive performance, and pain sensation. Modafinil is a stimulant drug marketed as a wakefulness and alertness promoting medication.

DETAILED DESCRIPTION:
The exact mechanism of action is unclear, and evidence has been gathered supporting a variety of different mechanisms including activity in a part of the brain that regulates wakefulness and alertness. The interaction between modafinil and alcohol has not been studied. The purpose of this study is to expand knowledge of the mood, memory, decision making, and pain relieving effects of each drug and how modafinil alters the effects of alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking adults who are 21 - 50 years of age.
2. Social or moderate drinkers who drink up to 14 drinks per week and are capable of drinking 3 drinks in a 90 minute time period.
3. Must have a Body Mass Index (BMI)>18 and <30.
4. If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or double barrier method [male condom, female condom, or diaphragm plus a spermicidal agent such as contraceptive foam, jelly or cream]).
5. Able and willing to provide written informed consent.
6. Able to understand and follow the instructions of the investigator, including all rating scales.
7. Develops temporary secondary hyperalgesia from the brief thermal sensitization stimulation procedure performed at the screening visit (Session 1).
8. Have a breath alcohol concentration (BAC) of 0.00 and a negative urine drug screen at all visits.

Exclusion Criteria:

1. Current or prior enrollment in an alcohol, or other drug treatment program or current legal problems relating to alcohol, or other drug use, including awaiting trial or supervision by a parole or probation officer.
2. Binge drinking more than once a week (>5 standard drinks in one session is a binge).
3. Currently trying to quit alcohol and/or "recreational" drug use.
4. Use of cocaine, amphetamines or other stimulants, hallucinogens, "ecstasy", or other psychoactive drugs, greater than 10 times in the last 24 months or at anytime in the past 60 days.
5. Positive for lifetime abnormal opioid use or prescription drug abuse.
6. Abusing inhalants (such as glue, toluene or other volatile substances), PCP, or ketamine greater than 10 times in the last 24 months, or at anytime in the past 60 days.
7. Use of caffeine or alcohol within 24 hours prior to the drug treatment sessions, or during study week except the alcohol supplied in the study. Heavy caffeine users who cannot tolerate stopping caffeine without symptoms are excluded.
8. Current tobacco users.
9. Use of any prescription medication (including topical), except birth control pills.
10. Use of any OTC medications during or 24 hours prior to study, including NSAIDS and "herbal" preparations (unless cleared by study physician). Exception is acetaminophen, which can be taken during the study period, but not within 12 hours prior or during the drug and alcohol study sessions 2-3.
11. Bilirubin or creatinine is more than 2 times the upper limit of normal range.
12. AST (SGOT), ALT (SGPT) or alkaline phosphatase is more than 2 ½ times the upper limit of normal range.
13. Positive urine drug screen or pregnancy test
14. Women of child bearing potential not currently using adequate means of contraception.
15. Coronary artery disease, uncontrolled hypertension, cardiac conduction abnormalities or significant arrhythmias, orthostatic mean blood pressure drop > than 25 mmHg, severe chronic obstructive pulmonary disease, or frequent headaches.
16. Any other clinically significant medical or psychiatric illness as determined by medical history, physical exam or screening blood tests, as judged by the study physician.
17. Chronic pain condition requiring regular physician visits and treatment under a physician's supervision.
18. Neurological dysfunction or psychiatric disorder severe enough to interfere with assessment of pain and sensory systems
19. Subjects receiving treatment with topical steroids (prescription or OTC) in areas to be stimulated.
20. Dermatopathology, skin hypersensitivity, or skin lesions in the area of measurements on the thigh and forearm.
21. Heat pain detection thresholds above 47°C/116.6°F on the arm.
22. Allergy to modafinil
23. Has received an investigational drug within 30 days prior to Study Visit 2.
24. Subjects who are unable to read or speak English.
25. Those, in the opinion of the investigator, who are considered unable to adhere to scheduled appointments, unlikely to comply with the study protocol, or who are unsuitable for any other reason.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-03; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Rowbotham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States